CLINICAL TRIAL: NCT03901573
Title: A Phase 1b/2a, Open Label Study to Evaluate Anti-tumor Efficacy and Safety of rhIL-7-hyFc (NT-I7) in Combination With Anti-PD-L1 (Atezolizumab) in Patients With Anti-PD-1/PD-L1 naïve or Relapsed/Refractory High-risk Skin Cancers
Brief Title: High-Risk Skin Cancers With Atezolizumab Plus NT-I7
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic decision by sponsor
Sponsor: NeoImmuneTech (Industry)
Collaborators: Immune Oncology Network (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIT-106; ION-02 (Other: Immune Oncology Network)
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Melanoma; Merkel Cell Carcinoma; Cutaneous Squamous Cell Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell | interventions — efineptakin alfa; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Checkpoint Inhibitor-Naive cSCC, MCC Pts (Experimental): Anti-PD-1/PD-L1 naïve patients with cSCC and MCC
  Interventions: Drug: NT-I7; Drug: atezolizumab
- Checkpoint Inhibitor-Relapsed/Refractory cSCC MCC Melanoma Pts (Experimental): Anti-PD-1/PD-L1 relapsed/refractory patients with cSCC, MCC and melanoma
  Interventions: Drug: NT-I7; Drug: atezolizumab

INTERVENTIONS:
Drug: NT-I7 — Dose Escalation (Phase 1b) - NT-I7 IM (intramuscular) on Day 1 of each Cycle until MTD or RP2D is achieved.
  Dose Expansion - NT-I7 IM (intramuscular) on Day 1 of each Cycle, at Maximum Tolerated Dose (MTD) or RP2D defined in escalation phase
  Other Names: efineptakin alfa; rhIL-7-hyFc
Drug: atezolizumab — Dose Escalation - atezolizumab IV (intravenous) on Day 1 of each Cycle
  Dose Expansion - atezolizumab IV (intravenous) on Day 1 of each Cycle
  Other Names: Tecentriq

SUMMARY:
The purpose of this study is to test whether the addition of NT-I7 to atezolizumab provides clinically meaningful outcomes for patients with anti-PD-1/PD-L1 naive or relapsed/refractory high-risk melanoma, Merkel Cell Carcinoma (MCC) and cutaneous Squamous Cell Carcinoma (cSCC)

DETAILED DESCRIPTION:
This is a Phase 1b/2a, open-label, multicenter study to evaluate the safety, tolerability and anti-tumor effect of NT-I7 (rhIL-7-hyFc) in combination with atezolizumab (MPDL3280A, anti-PD-L1) in patients with anti-PD-1/PD-L1 naïve or relapsed/refractory high-risk skin cancers including cutaneous Squamous Cell Carcinoma (cSCC), Merkel Cell Carcinoma (MCC) and melanoma.

This study has been designed to evaluate the safety and tolerability, including the Maximum Tolerated Dose (MTD) or recommended Phase 2 dose (RP2D), of NT-I7 in combination with atezolizumab.

There are two phases to this study:

* Phase 1b, a NT-I7 dose-escalation phase to determine the MTD or RP2D
* Phase 2a, a non-randomized parallel dose expansion phase to confirm the MTD or RP2D in both arms.

Arm I: Anti-PD-1/PD-L1 (checkpoint inhibitors, CPI) naïve patients with cSCC and MCC

Arm II: Anti-PD-1/PD-L1 relapsed/refractory patients with cSCC, MCC and melanoma

Number of Patients A total of up to 84 patients will be enrolled; Up to 24 patients will be enrolled in the Phase 1b (up to 6 patients per dose level, using 3 + 3 design), and 60 patients will be enrolled in the Phase 2a (24 patients in Arm I, i.e., 12 patients for each indication, and 36 in Arm II, i.e., 12 patients for each indication).

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients must be ≥18 years of age on day of signing informed consent document.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%).
3. Patients must have adequate organ and marrow function.
4. Patients positive for HIV can be considered.
5. Arm I - cSCC: Patients must have biopsy-proven metastatic cSCC or locoregional cSCC that has recurred following standard locoregional therapy with surgery and/or radiation therapy; MCC: Patients must have biopsy-proven metastatic MCC or locoregional MCC in need of systemic therapy, including patients that have not had prior systemic therapy or have recurred following standard locoregional therapy with surgery and/or radiation therapy. Prior chemotherapy is allowed.
6. Arm II - MCC: Patients must have biopsy-proven metastatic MCC or locoregional MCC that has recurred following anti-PD-1 or anti-PD-L1, or has SD following anti-PD-1 or anti-PD-L1, defined as 12 weeks of SD per RECIST 1.1; cSCC: Patients must have biopsy-proven metastatic cSCC or locoregional cSCC that has recurred following anti-PD-1 or anti-PD-L1, or has SD following anti-PD-1 or anti-PD-L1, defined as 12 weeks of SD per RECIST 1.1; Melanoma: Patients must have biopsy-proven metastatic melanoma or locoregional melanoma that has recurred following anti-PD-1, anti-PD-L1, or has SD following anti-PD-1 or anti-PD-L1, defined as 12 weeks of SD per RECIST 1.1.

Note: Prior therapy with ipilimumab is allowed (subject to a 6-week washout period) but not required.

Note: Progression following targeted therapies (e.g., BRAF inhibitor and/or MEK inhibitor) or other approved (e.g., talimogene laherparepvec [T-VEC]) or investigational therapies is allowed.

Key Exclusion Criteria:

1. Pregnancy, lactation, or breastfeeding.
2. Significant cardiovascular disease.
3. Poorly controlled Type 2 diabetes mellitus.
4. Major surgical procedure, other than for diagnosis, within 28 days prior to Cycle 1, Day 1, or anticipation of need for a major surgical procedure during the study.
5. Patients who have had chemotherapy or radiotherapy within 2 weeks (4 weeks for nitrosoureas or systemic mitomycin C) prior to Cycle 1, Day 1.
6. Patients who had prior treatment with immune CPIs, immunomodulatory monoclonal antibodies (mAbs), and/or mAb-derived therapies within 6 weeks before the initiation of study treatment, except for prior anti-PD-L1/anti-PD-1, which requires a 3-week washout period.
7. Patients who have received treatment with any other investigational agent within 4 weeks prior to Cycle 1, Day 1.
8. Patients who have received treatment and failed therapy with checkpoint inhibition plus a T-cell growth factor, e.g., IL-2 (NTKR-204), IL-15 (ALT-803) or IL-7 (CYT107).
9. Patients with known primary central nervous system (CNS) malignancy, untreated CNS metastases, or active CNS metastases (progressing or requiring corticosteroids for symptomatic control) are excluded, with some exceptions.
10. Patients who have leptomeningeal disease.
11. Patients with autoimmune disease history.
12. Patients who have received treatment with systemic immunosuppressive medications within 2 weeks prior to Cycle 1, Day 1.
13. Patients who have a history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
14. Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening).
15. Patients with active tuberculosis (TB).
16. Patients who have severe infections within 4 weeks prior to Cycle 1, Day 1.
17. Patients who have signs or symptoms of recent infection (not meeting the above criteria for severe infections) within 2 weeks before initiation of study treatment.
18. Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.
19. Patients who have received a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1 or anticipate that such a live attenuated vaccine be required during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NgocDiep Le, MD, PhD, Study Chair — NeoImmuneTech; Martin Cheever, MD, Study Director — Fred Hutchinson Cancer Center; Brian Gastman, MD, Principal Investigator — The Cleveland Clinic
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Northwestern University, Chicago, Illinois
  - Dana Farber, Boston, Massachusetts
  - MGH, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Mt Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b-Dose Level 1: NT-I7 120 µg/kg IM Q3W
  + atezolizumab 1200 mg IV Q3W
- Phase 1b-Dose Level 2: NT-I7 360 µg/kg IM Q3W
  + atezolizumab 1200 mg IV Q3W
- Phase 1b-Dose Level 3: NT-I7 840 µg/kg IM Q3W
  + atezolizumab 1200 mg IV Q6W
- Phase 1b-Dose Level 4; Phase 2-: NT-I7 1200 µg/kg IM Q6W
  + atezolizumab 1200 mg IV Q6W
Period: Overall Study
Arm/Group | Phase 1b-Dose Level 1 | Phase 1b-Dose Level 2 | Phase 1b-Dose Level 3 | Phase 1b-Dose Level 4 | Phase 2-
Started | 3 | 3 | 7 | 3 | 15
Completed | 2 | 2 | 4 | 3 | 7
Not Completed | 1 | 1 | 3 | 0 | 8

BASELINE CHARACTERISTICS:
Population: The study enrolled 16 subjects in Phase 1b and 15 subjects in Phase 2a, all of whom received treatment. The Arm/Group has been combined based on the dosing regimen of NT-I7 per study design: Phase 1b, DL1-3 every 3 weeks (Q3W); Phase 1b DL4 and Phase 2a, Q6W.
Groups:
- Phase 1b; Phase 2a: Baseline characteristics are summarized by dose level (Phase 1b: 120, 360, 840, 1200 μg/kg; Phase 2a: 1200 μg/kg) rather than by Arm because pooling was pre-specified in the Statistical Analysis Plan (Section 4.2.1) and protocol. Efficacy analyses also pool Phase 1b doses (120-840 μg/kg) and Phase 2a 1200 μg/kg dose. This approach reflects study design and planned analyses.
- Total: Total of all reporting groups
Arm/Group | Phase 1b | Phase 2a | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 9 | 11 | 20
Age, Continuous [Median (Full Range); unit: years] | 65.4 [46 to 82] | 65.7 [39 to 82] | 65.58 [39 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Weight [Median (Full Range); unit: kg] | 81.42 [58.3 to 123.4] | 78.00 [54.3 to 111] | 79.71 [54.3 to 123.4]

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: To Evaluate the Safety and Tolerability of NT-I7 in Combination With Atezolizumab, Including Estimation of the Maximum Tolerated Dose and/or the Recommended Phase 2 Dose
Description: 1. Incidence, nature, and severity of adverse events graded according to NCI CTCAE 5.0
  2. Incidence and nature of dose-limiting toxicities (DLTs)
  Note: ORR (Defined as the percentage of patients who have at least one confirmed partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1). ORR is included in Phase 2a Primary Outcome Measure.
Time Frame: 1. On or after administration of study treatment through 30 days after the last dose of study treatment (approximately 25 months after enrollment) 2.First 21 days (C1/D1 through Day 21)
Population: Safety: All patients who receive at least 1 dose of the investigational regimen ; DLT: All patients who receive at least 1 dose of the investigational regimen and complete the full 3-week DLT window or who do not complete the full 3-week DLT window due to the occurrence of a DLT.; Analyses of adverse events will be performed for those events that are considered treatment emergent.(Subjects with one or more AEs within a level of MedDRA are counted only once in that level)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b-Dose Level 1 | Phase 1b-Dose Level 2 | Phase 1b-Dose Level 3 | Phase 1b-Dose Level 4 | Phase 2-
Number analyzed (Participants) | 3 | 3 | 7 | 3 | 15
Participants
  Incidence of Treatment-Related TEAE | 3 | 3 | 7 | 3 | 14
  Patient Incidence of Serious Treatment-Emergent Adverse Events | 1 | 0 | 5 | 1 | 9
  Patient Incidence of Serious Treatment-Related Adverse Events | 0 | 0 | 3 | 0 | 4
  Patient Incidence of Adverse Events of Special Interest | 2 | 1 | 3 | 0 | 9
  Experienced a DLT | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Phase 2a: To Evaluate the Objective Response Rate (ORR) According to RECIST 1.1 and iRECIST, as Determined by the Investigator
Description: Pooling of dose levels for this Outcome Measure was pre-specified in the Statistical Analysis Plan (SAP Section 4.2.1) and the study protocol. Phase 1b dose-escalation results are summarized by dose level (120, 360, 840, 1200 µg/kg), and Phase 2a results under 1200 µg/kg. Efficacy analyses pool Phase 1b doses (120-840 µg/kg) and the Phase 2a 1200 µg/kg dose to reflect the predefined analysis strategy and study objectives. This approach was chosen due to small sample sizes and early study termination, as documented in the Clinical Study Report (CSR).
Time Frame: C1D1 until the start of a new anticancer treatment, disease progression, pregnancy, death, withdrawal of consent or end of study, whichever occurs first, up to 1 year
Population: The Arm/Group has been categorized based on the dosing regimen of NT-I7 per study design: Phase 1b, DL1-3 every 3 weeks (Q3W); Phase 1b DL4 and Phase 2a, Q6W.treatment and have at least one evaluable post baseline tumor assessment.
Measure: Count of Participants; unit: Participants
Groups:
- NT-I7 Dose Levels + Atezolizumab (120-840 µg/kg): NT-I7 Dose Levels (120-840 µg/kg) + Atezolizumab 1200 mg. Consisted of all subjects that were enrolled in Cohort 1 NT-I7 120µg/kg, Cohort 2 NT-I7 840µg/kg and Cohort 3 NT-I7 Dose Levels 840 µg/kg
- NT-I7 Dose Levels + Atezolizumab (1200 µg/kg): NT-I7 Dose Levels (1200 µg/kg) + Atezolizumab 1200mg. Consisted of all subjects in cohort 4 NT-I7 Dose Levels (1200 µg/kg) and Phase 2a RP2D NT-I7 Dose Levels (1200 µg/kg)
Arm/Group | NT-I7 Dose Levels + Atezolizumab (120-840 µg/kg) | NT-I7 Dose Levels + Atezolizumab (1200 µg/kg)
Number analyzed (Participants) | 12 | 15
Participants
  Complete response | 0 | 0
  Partial response | 0 | 2
  Stable disease | 9 | 6
  Progressive disease | 3 | 7

3. Secondary Outcome: To Evaluate Immunogenicity of NT-I7 in Combination With Atezolizumab
Description: The ADA status will be defined using the baseline and postbaseline results. Anti-drug antibody negative is defined as negative results at all time points. Anti-drug antibody positive is defined as a positive result at any time point, including baseline.
Time Frame: C1D1 through end of 90-day follow-up
Population: All patients who receive at least 1 dose of the investigational regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b-Dose Level 1 | Phase 1b-Dose Level 2 | Phase 1b-Dose Level 3 | Phase 1b-Dose Level 4 | Phase 2-
Number analyzed (Participants) | 3 | 3 | 7 | 3 | 15
Participants
  Baseline: Subjects that are ADA Positive | 0 | 0 | 0 | 0 | 1
  Baseline: Subjects that are ADA Negative | 3 | 3 | 7 | 3 | 12
  Baseline: n (Missing) | 0 | 0 | 0 | 0 | 2
  C2D1: Subjects that are ADA Negative | 0 | 1 | 4 | 0 | 2
  C2D1: Subjects that are ADA Positive | 3 | 2 | 2 | 3 | 11
  C2D1: n (Missing) | 0 | 0 | 1 | 0 | 2
  End of Treatment: Subjects that are ADA Negative | 0 | 0 | 0 | 0 | 0
  End of Treatment: n (Missing) | 0 | 1 | 0 | 0 | 6
  End of Treatment: Subjects that are ADA Positive | 3 | 2 | 7 | 3 | 9
  90-Day Follow up: Subjects that are ADA Positive | 2 | 2 | 4 | 3 | 4
  90-Day Follow up: n (Missing) | 1 | 1 | 3 | 0 | 11
  90-Day Follow up: Subjects that are ADA Negative | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: To Make a Preliminary Assessment of the Anti-tumor Activity of NT-I7 in Combination With Atezolizumab
Description: Pooling of dose levels for this Outcome Measure was also pre-specified in the SAP and study protocol to maintain consistency across efficacy endpoints. For this Outcome Measure (e.g., Disease Control Rate), pooled groups were defined as Phase 1b (120-840 µg/kg) and Phase 2a (1200 µg/kg). This approach aligns with the predefined analyses and study objectives and prevents misleading subgroup estimates given the limited enrollment and early study termination.
Time Frame: as for outcome 2
Population: Defined as the time from the first occurrence of stable disease or better (PR or CR or SD) to the time of the first documented disease progression or death from any cause, whichever occurs first per RECIST v1.1. The Arm/Group has been categorized based on the dosing regimen of NT-I7 per study design: Phase 1b, DL1-3 every 3 weeks (Q3W); Phase 1b DL4 and Phase 2a, Q6W.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- NT-I7 Dose Levels (NT-I7 120-840 µg/kg) + Atezolizumab: NT-I7 Dose Levels (120-840 µg/kg) + Atezolizumab 1200 mg. Consisted of all subjects that were enrolled in Cohort 1 NT-I7 120µg/kg, Cohort 2 NT-I7 840µg/kg and Cohort 3 NT-I7 Dose Levels 840 µg/kg
- NT-I7 Dose Levels (1200 µg/kg) + Atezolizumab: NT-I7 Dose Levels (1200 µg/kg) + Atezolizumab 1200mg. Consisted of all subjects in cohort 4 NT-I7 Dose Levels (1200 µg/kg) and Phase 2a RP2D NT-I7 Dose Levels (1200 µg/kg)
Arm/Group | NT-I7 Dose Levels (NT-I7 120-840 µg/kg) + Atezolizumab | NT-I7 Dose Levels (1200 µg/kg) + Atezolizumab
Number analyzed (Participants) | 12 | 15
Months
  Duration of stable disease | 2.2 [1.41 to 12.25] | 2.0 [1.45 to 2.27]
  Progression -Free Survival, RECIST 1.1 | 4.2 [2.07 to 6.93] | 3.5 [1.87 to 4.24]
  Overall Survival | 11.1 [3.81 to 22.24] | NA [5.06 to NA] — The cohort didn't reach 50% survival within the observation period

5. Secondary Outcome: To Make a Preliminary Assessment of the Anti-tumor Activity of NT-I7 in Combination With Atezolizumab (DCR)
Description: For Outcome Measure 4 and 5, pooling was also pre-specified in SAP Section 4.8 and CSR Section 11.4. Kaplan-Meier analyses were conducted on pooled groups for interpretability and statistical validity. Separate reporting by Arm was not feasible due to small sample sizes and early termination.
Time Frame: as for outcome 2
Population: All patients who received at least one cycle of study treatment and have at least one evaluable post baseline tumor assessment. The Arm/Group has been categorized based on the dosing regimen of NT-I7 per study design: Phase 1b, DL1-3 every 3 weeks (Q3W); Phase 1b DL4 and Phase 2a, Q6W.
Measure: Number; unit: percentage of participants
Arm/Group | NT-I7 Dose Levels (NT-I7 120-840 µg/kg) + Atezolizumab | NT-I7 Dose Levels (1200 µg/kg) + Atezolizumab
Number analyzed (Participants) | 12 | 15
percentage of participants | 75.0 | 53.3

ADVERSE EVENTS:
Time Frame: On or after administration of study treatment through 30 days after the last dose of study treatment (approximately 25 months after enrollment)
Description: Incidence of Treatment-Related TEAE by MedDRA System Organ Class and Preferred Term (Safety Population)
Arm/Group | Phase 1b-Dose Level 1 | Phase 1b-Dose Level 2 | Phase 1b-Dose Level 3 | Phase 1b-Dose Level 4 | Phase 2-
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/3 | 5/7 | 1/3 | 8/15
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 5/7 | 1/3 | 9/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 3/3 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b-Dose Level 1 (N=3) | Phase 1b-Dose Level 2 (N=3) | Phase 1b-Dose Level 3 (N=7) | Phase 1b-Dose Level 4 (N=3) | Phase 2- (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Loss of personal independence in daily activities (Social circumstances) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b-Dose Level 1 (N=3) | Phase 1b-Dose Level 2 (N=3) | Phase 1b-Dose Level 3 (N=7) | Phase 1b-Dose Level 4 (N=3) | Phase 2- (N=15)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0
Dry eye (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 1
Blood lactate dehydrogenase (Investigations) | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2 | 0 | 2
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 2
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 3 | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 1 | 1 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 (0) | 2 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 3
Hypophosphatasemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Pain in extremity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 2 | 3
Confusional state (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 3
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 4 | 2 | 8
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 0 | 4
Injection site dryness (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 1 | 3 | 2 | 7
Localized oedema (General disorders) | 0 | 0 | 1 | 0 | 1
Nodule (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 5
Oedema peripheral (General disorders) | 1 | 1 | 2 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Hip fracture (Investigations) | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 1 | 0
Enterobacter test positive (Investigations) | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1
Investigation abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Lymphocyte count (Investigations) | 0 | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1
Respiratory rate increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Hypermagnesaemi (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Loss of personal independence in daily activities (Social circumstances) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Troponin T increased (Investigations) | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03901573/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03901573/SAP_001.pdf
  • Informed Consent Form: Main (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03901573/ICF_002.pdf
  • Informed Consent Form: Addendum (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03901573/ICF_003.pdf